CLINICAL TRIAL: NCT00112242
Title: Vaccination of Patients With Stage III or IV Malignant Melanoma With Melanoma Antigen Peptides [Melan-A/Mart-1 Analog (ELA), NY-ESO-1b(A) Analog and MAGE-A10] and Montanide Adjuvant
Brief Title: Immunotherapy of Stage III/IV Melanoma Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Collaborators: Ludwig Institute for Cancer Research (Other)
Responsible Party: Principal Investigator, Prof Olivier Michielin, M.D., Ph.D., Professor, Centre Hospitalier Universitaire Vaudois
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LUD 2001-003
Record Dates: First submitted 2005-05-31; First posted 2005-06-01 (Estimated); Results first posted 2020-06-18 (Actual); Last update posted 2020-06-18 (Actual); Status verified 2020-06

CONDITIONS: Melanoma
Keywords: Immunotherapy; Vaccination; Melanoma; Melan-A/Mart-1 peptide; MAGE-A10 peptide; NY-ESO-1 peptide; Montanide; CpG
MeSH Terms: conditions — Melanoma | interventions — MART-1 Antigen; Monatide (IMS 3015); MAGE-A10 antigen; cytidylyl-3'-5'-guanosine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- 1. Melan-A ELA (Experimental): 500 mcg Melan-A ELA analog peptide + 1 ml Montanide ISA-51
  Interventions: Biological: Melan-A ELA + Montanide
- 2. Melan-A ELA + NY-ESO-1b + MAGE-A10 (Experimental): 500 mcg Melan-A ELA analog peptide + 500 mcg NY-ESO-1b(A) analog peptide + 500 mcg MAGE-A10 peptide + 1 ml Montanide ISA-51
  Interventions: Biological: Melan-A ELA + NY-ESO-1b + MAGE-A10 + Montanide
- 3. Melan-A ELA + NY-ESO-1b + MAGE-A10 + CpG (Experimental): 500 mcg Melan-A ELA analog peptide + 500 mcg NY-ESO-1b(A) analog peptide + 500 mcg MAGE-A10 peptide + 1 ml Montanide ISA-51 + 2.5 mg CpG-7909/PF-3512676
  Interventions: Biological: Melan-A -ELA + NY-ESO-1b + MAGE-A10 peptide + Montanide + CpG
- 4. Melan-A EAA/ELA + NY-ESO-1lp + MAGE-A10+ CpG (Experimental): * If patient is HLA-A2 positive: 100 mcg Melan-A EAA native peptide (during first cycle) or 100 mcg ELA analog peptide (during other cycles) + 500 mcg NY-ESO-1lp long peptide + 100 mcg MAGE-A10 peptide + 1 ml Montanide ISA-51 (no Montanide during cycle 3) + 2.5 mg CpG-7909/PF-3512676
  * If patient is HLA-A2 negative: 500 mcg NY-ESO-1lp long peptide+ 1 ml Montanide ISA-51 (no Montanide during cycle 3) + 2.5 mg CpG-7909/PF-3512676
  Interventions: Biological: Melan-A-EAA/ELA + NY-ESO-1 lp + MAGE-A10 + Montanide + CpG
- 5. Melan-A EAA/ELA + NY-ESO-1lp + MAGE-A10+ CpG+ IL-2 (Experimental): * If patient is HLA-A2 positive: 100 mcg Melan-A EAA native peptide (during first cycle) or 100 mcg ELA analog peptide (during other cycles) + 500 mcg NY-ESO-1lp long peptide + 100 mcg MAGE-A10 peptide + 1 ml Montanide ISA-51 (no Montanide during cycle 3) + 2.5 mg CpG-7909/PF-3512676 + low dose IL-2
  * If patient is HLA-A2 negative: 500 mcg NY-ESO-1lp long peptide+ 1 ml Montanide ISA-51 (no Montanide during cycle 3) + 2.5 mg CpG-7909/PF-3512676 + low dose IL-2
  Interventions: Biological: Melan-A-EAA/ELA + NY-ESO-1 lp + MAGE-A10 + Montanide + CpG+ IL-2

INTERVENTIONS:
Biological: Melan-A ELA + Montanide — A maximum of 3 vaccination cycles (cycles 1-3) has been given, each cycle consisting of 4 vaccines in 4 week intervals. The intervals between cycles were 8 weeks. After 3 cycles, patients without major tumor progression requiring other treatment who showed an immunological response received "booster vaccinations" every 3 months.
  Arms: 1. Melan-A ELA
Biological: Melan-A ELA + NY-ESO-1b + MAGE-A10 + Montanide — A maximum of 3 vaccination cycles (cycles 1-3) has been given, each cycle consisting of 4 vaccines in 4 week intervals. The intervals between cycles were 8 weeks. After 3 cycles, patients without major tumor progression requiring other treatment who showed an immunological response received "booster vaccinations" every 3 months.
  Arms: 2. Melan-A ELA + NY-ESO-1b + MAGE-A10
Biological: Melan-A -ELA + NY-ESO-1b + MAGE-A10 peptide + Montanide + CpG — A maximum of 3 vaccination cycles (cycles 1-3) has been given, each cycle consisting of 4 vaccines in 4 week intervals. The intervals between cycles were 8 weeks. After 3 cycles, patients without major tumor progression requiring other treatment who showed an immunological response received "booster vaccinations" every 3 months.
  Arms: 3. Melan-A ELA + NY-ESO-1b + MAGE-A10 + CpG
Biological: Melan-A-EAA/ELA + NY-ESO-1 lp + MAGE-A10 + Montanide + CpG — A maximum of 3 vaccination cycles (cycles 1-3) has been given, each cycle consisting of 4 vaccines in 4 week intervals. The intervals between cycles were 8 weeks. After 3 cycles, patients without major tumor progression requiring other treatment who showed an immunological response received "booster vaccinations" every 3 months.
  Arms: 4. Melan-A EAA/ELA + NY-ESO-1lp + MAGE-A10+ CpG
Biological: Melan-A-EAA/ELA + NY-ESO-1 lp + MAGE-A10 + Montanide + CpG+ IL-2 — A maximum of 3 vaccination cycles (cycles 1-3) has been given, each cycle consisting of 4 vaccines in 4 week intervals. The intervals between cycles were 8 weeks. After 3 cycles, patients without major tumor progression requiring other treatment who showed an immunological response received "booster vaccinations" every 3 months.
  Arms: 5. Melan-A EAA/ELA + NY-ESO-1lp + MAGE-A10+ CpG+ IL-2

SUMMARY:
The purpose of this study is to determine whether vaccination with melanoma antigen peptides [Melan-A/Mart-1 (both EAA and ELA), NY-ESO-1b analog, Long NY-ESO-1 LP and MAGE-A10] and Montanide, CpG adjuvants and low dose rIL-2 can induce an immune response in melanoma patients and to assess the safety of this vaccination.

DETAILED DESCRIPTION:
Current peptide vaccines suffer from low efficiency, since they induce only weak immune activation. We have recently confirmed that in humans the immune response was readily detectable in local lymph nodes while no or only weak activation could be identified in circulating lymphocytes. Increased doses of antigen and adjuvant allow a better extension from local to systemic immune responses.

* Group 1 : vaccination with Melan-A analog (ELA) peptide + Montanide
* Group 2 : vaccination with Melan-A analog (ELA), NY-ESO-1b analog and MAGE-A10 peptides + Montanide
* Group 3: vaccination with Melan-A analog (both EAA and ELA), Mage-A10, NY-ESO-1 peptides+ Montanide + CpG adjuvant
* Group 4: vaccination with Melan-A (ELA), Mage-A10,long NY-ESO-1LP peptides + Montanide + CpG
* Group 5: vaccination with Melan-A (both EAA and ELA), Mage-A10, long NY-ESO-1 LP peptides + Montanide + CpG + low dose rIL-2

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed stage III or stage IV melanoma with at least one metastatic lymph node and/or at least one in-transit metastasis. According to the AJCC rules, this includes all patients with stage IV and stage III. Patients with or without measurable disease may be included.
2. Tumor expression of Melan-A by reverse transcriptase and polymerase chain reaction (RT-PCR) analysis for patients of group I.

   Tumor expression of Melan-A and at least one of the tumor antigens MAGE-A10, NY-ESO-1, or LAGE-1 by rt-PCR analysis for patients of group II and III and for HLA-A2+ patients of groups IV and V. HLA-A2 negative patients of groups IV and V must only have NY-ESO-1 positive tumors to be eligible, while expression of Melan-A and MAGE-A10 is unimportant.

   If no frozen tissue is available, immunohistochemistry may be performed to detect tumor expression of Melan-A and NY-ESO-1.
3. HLA-A2 positive (serological or molecular typing of Peripheral Blood Lymphocytes (PBL) for patients of groups 1 to 3. Patients of groups 4 and 5 may either be HLA-A2+ or HLA-A2-.
4. Expected survival of at least five months.
5. Full recovery from surgery.
6. Karnofsky scale performance status of 70% or more.
7. The following laboratory results:

   Neutrophil count sup or equal 2.0 x 10^9/L Lymphocyte count sup or equal 0.5 x 10^9/L Platelet count sup or equal 100 x 10^9/L Creatinine ≤ 2 mg/dL (180 micromol/L) Bilirubin ≤ 2mg/dL (34 micromol/L) Granulocyte count > 2.5x10^9/L AST < 2x upper limit of normal aPTT: within the normal ranges of the laboratory ± 25 %
8. Age > 18 years.
9. Able to give written informed consent.

Exclusion Criteria:

1. Clinically significant heart disease (NYHA Class III or IV).
2. Other serious illnesses, e.g., serious infections requiring antibiotics, uncontrolled peptic ulcer, or central nervous system disorders with major dysfunction.
3. History of immunodeficiency disease or autoimmune disease.
4. Known HIV positivity.
5. Known seropositivity for hepatitis B surface antigen.
6. Chemotherapy, radiation therapy, or immunotherapy within 4 weeks before study entry (6 weeks for nitrosoureas).
7. Concomitant treatment with steroids, antihistamine drugs. Topical or inhalational steroids are permitted.
8. Participation in any other clinical trial involving another investigational agent within 4 weeks prior to enrollment.
9. Pregnancy or lactation.
10. Women of childbearing potential not using a medically acceptable means of contraception.
11. Psychiatric or addictive disorders that may compromise the ability to give informed consent.
12. Lack of availability of the patient for immunological and clinical follow-up assessment.
13. Coagulation or bleeding disorders.
14. Metastatic disease to the central nervous system, unless treated and stable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2004-02; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Michielin, MD PhD, Principal Investigator — Lausanne University Hospital (Centre Hospitalier Universitaire Vaudois)
Locations (2):
- Switzerland (2):
  - Oncology Department, Lausanne University Hospital (CHUV) and University of Lausanne, Lausanne, Canton of Vaud
  - Division of Oncology at the Geneva University Hospital, Geneva

REFERENCES:
- [Result] Baumgaertner P, Costa Nunes C, Cachot A, Maby-El Hajjami H, Cagnon L, Braun M, Derre L, Rivals JP, Rimoldi D, Gnjatic S, Abed Maillard S, Marcos Mondejar P, Protti MP, Romano E, Michielin O, Romero P, Speiser DE, Jandus C. Vaccination of stage III/IV melanoma patients with long NY-ESO-1 peptide and CpG-B elicits robust CD8+ and CD4+ T-cell responses with multiple specificities including a novel DR7-restricted epitope. Oncoimmunology. 2016 Sep 9;5(10):e1216290. doi: 10.1080/2162402X.2016.1216290. eCollection 2016. PMID 27853637
- [Result] Hebeisen M, Schmidt J, Guillaume P, Baumgaertner P, Speiser DE, Luescher I, Rufer N. Identification of Rare High-Avidity, Tumor-Reactive CD8+ T Cells by Monomeric TCR-Ligand Off-Rates Measurements on Living Cells. Cancer Res. 2015 May 15;75(10):1983-91. doi: 10.1158/0008-5472.CAN-14-3516. Epub 2015 Mar 25. PMID 25808864
- [Result] Bordry N, Costa-Nunes CM, Cagnon L, Gannon PO, Abed-Maillard S, Baumgaertner P, Murray T, Letovanec I, Lazor R, Bouchaab H, Rufer N, Romano E, Michielin O, Speiser DE. Pulmonary sarcoid-like granulomatosis after multiple vaccinations of a long-term surviving patient with metastatic melanoma. Cancer Immunol Res. 2014 Dec;2(12):1148-53. doi: 10.1158/2326-6066.CIR-14-0143. Epub 2014 Oct 2. PMID 25277238
- [Derived] Costa-Nunes C, Cachot A, Bobisse S, Arnaud M, Genolet R, Baumgaertner P, Speiser DE, Sousa Alves PM, Sandoval F, Adotevi O, Reith W, Protti MP, Coukos G, Harari A, Romero P, Jandus C. High-throughput Screening of Human Tumor Antigen-specific CD4 T Cells, Including Neoantigen-reactive T Cells. Clin Cancer Res. 2019 Jul 15;25(14):4320-4331. doi: 10.1158/1078-0432.CCR-18-1356. Epub 2019 Apr 23. PMID 31015344

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were screened and enrolled at 2 sites in Switzerland, the CHUV in Lausanne and the HUG in Geneva.
Pre-assignment Details: The assignment to a group was done according to tumor antigen (i.e., Melan-A, MAGE-A10, NY-ESO-1b[A]) and HLA expression (HLA-A2).
Groups:
- 1. Melan-A ELA: 500 mcg Melan-A ELA analog peptide + 1 ml Montanide
- 2. Melan-A ELA + NY-ESO-1b(A) + MAGE-A10: 500 mcg Melan-A ELA analog peptide + 500 mcg NY-ESO-1b(A) analog peptide + 500 mcg MAGE-A10 peptide + 1 ml Montanide
- 3. Melan-A ELA + NY-ESO-1b(A) + MAGE-A10 + CpG: 500 mcg Melan-A ELA analog peptide + 500 mcg NY-ESO-1b(A) analog peptide + 500 mcg MAGE-A10 peptide + 1 ml Montanide + 2.5 mg CpG-7909/PF-3512676
- 4. Melan-A EAA/ELA + NY-ESO-1lp + MAGE-A10+ CpG: * If patient is HLA-A2 positive: 100 mcg Melan-A EAA native peptide (during first cycle) or 100 mcg ELA analog peptide (during other cycles) + 500 mcg NY-ESO-1lp long peptide + 100 mcg MAGE-A10 peptide + 1 ml Montanide (no Montanide during cycle 3) + 2.5 mg CpG-7909/PF-3512676
  * If patient is HLA-A2 negative: 500 mcg NY-ESO-1lp long peptide+ 1 ml Montanide (no Montanide during cycle 3) + 2.5 mg CpG-7909/PF-3512676
- 5. Melan-A EAA/ELA + NY-ESO-1lp + MAGE-A10+ CpG + IL-2: * If patient is HLA-A2 positive: 100 mcg Melan-A EAA native peptide (during first cycle) or 100 mcg ELA analog peptide (during other cycles) + 500 mcg NY-ESO-1lp long peptide + 100 mcg MAGE-A10 peptide + 1 ml Montanide (no Montanide during cycle 3) + 2.5 mg CpG-7909/PF-3512676 + low dose IL-2
  * If patient is HLA-A2 negative: 500 mcg NY-ESO-1lp long peptide+ 1 ml Montanide (no Montanide during cycle 3) + 2.5 mg CpG-7909/PF-3512676 + low dose IL-2
Period: Overall Study
Arm/Group | 1. Melan-A ELA | 2. Melan-A ELA + NY-ESO-1b(A) + MAGE-A10 | 3. Melan-A ELA + NY-ESO-1b(A) + MAGE-A10 + CpG | 4. Melan-A EAA/ELA + NY-ESO-1lp + MAGE-A10+ CpG | 5. Melan-A EAA/ELA + NY-ESO-1lp + MAGE-A10+ CpG + IL-2
Started | 10 | 5 | 5 | 10 | 9 (One patient received only 1 vaccine however this minimum dose allowed the safety evaluation)
Cycle 1 Completed | 10 | 5 | 5 | 9 | 7
Cycle 2 Completed | 8 | 3 | 4 | 8 | 4
Cycle 3 Completed | 5 | 3 | 4 | 4 | 2
Completed (Received 3 cycles of treatment) | 5 | 3 | 4 | 4 | 2
Not Completed | 5 | 2 | 1 | 6 | 7

BASELINE CHARACTERISTICS:
Population: At study entry the melanoma antigens expression and HLA expression analysis was done in order to know at what group of treatment the patient had to be assigned
Groups:
- Single Peptide Vaccination: Montanide + Melan-A analogue peptide
  Montanide + Melan-A analogue peptide: 1 ml Montanide+ 500 mcg Melan-A analog peptide
- Peptide Combination Vaccination: Montanide + Melan-A analog peptide + NY-ESO-1 analog peptide + Mage10 peptide
  Montanide + Melan-A analog peptide + NY-ESO-1 analog peptide + Mage10 peptide: 1 ml Montanide + 500 mcg Melan-A analog peptide + 500 mcg NY-ESO-1 analog peptide + 500 mcg Mage10 peptide
- Peptide Combination Vaccination + CpG: Montanide + CpG-7909/PF-3512676+Melan-A analog peptide + NY-ESO-1 analog peptide + Mage10 peptide
  Montanide + CpG-7909 / PF-3512676+Melan-A analog peptide + NY-ESO-1 analog peptide + Mage10 peptide: 1 ml Montanide + 2.5 mg CpG-7909/PF-3512676 + 500 mcg Melan-A analog peptide, 500 mcg + NY-ESO-1 analog peptide + 500 mcg Mage10 peptide
- Native and Analog Peptide Combination Vaccination + CpG: Montanide + CpG-7909/PF-3512676 + Melan-A native and analog peptides + NY-ESO-1 long peptide + Mage10 peptide
  Montanide + CpG-7909/PF-3512676 + Melan-A native and analog peptides + NY-ESO-1 long peptide + Mage10 peptide: 1 ml Montanide + 2.5 mg CpG-7909/PF-3512676 + 100 mcg Melan-A native and analog peptides + 500 mcg NY-ESO-1 long peptide + 100 mcg Mage10 peptide
- Native and Analog Peptide Combination Vaccination + CpG + IL-2: Montanide + CpG-7909/PF-3512676 + Melan-A native and analog peptides + NY-ESO-1 long peptide + Mage10 peptide + low dose IL-2
  Montanide + CpG-7909/PF-3512676 + Melan-A native and analog peptides + NY-ESO-1 long peptide + Mage10 peptide + low dose IL-2: 1 ml Montanide + 2.5 mg CpG-7909/PF-3512676 + 100 mcg Melan-A native and analog peptides + 500 mcg NY-ESO-1 long peptide + 100 mcg Mage10 peptide + low dose IL-2
- Total: Total of all reporting groups
Arm/Group | Single Peptide Vaccination | Peptide Combination Vaccination | Peptide Combination Vaccination + CpG | Native and Analog Peptide Combination Vaccination + CpG | Native and Analog Peptide Combination Vaccination + CpG + IL-2 | Total
Number analyzed (Participants) | 10 | 5 | 5 | 10 | 8 | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 3 | 3 | 8 | 6 | 26
  >=65 years | 4 | 2 | 2 | 2 | 2 | 12
Age, Continuous [Median (Full Range); unit: years] | 61.8 [34.1 to 77.1] | 58.8 [37.8 to 73.8] | 64.9 [47.3 to 78.1] | 59.9 [31.4 to 65.5] | 59.2 [35.6 to 66.6] | 60.1 [31.4 to 78.1]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 2 | 2 | 3 | 12
  Male | 7 | 3 | 3 | 8 | 5 | 26
Region of Enrollment [Count of Participants; unit: Participants]
  Switzerland | 10 | 5 | 5 | 10 | 8 | 38

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean Number of Adverse Events (Serious and Non Serious Events)
Description: Safety of the vaccination was assessed according to the National Cancer Institute Common Toxicity Criteria (NCI CTC) scale. The adverse events (AE) and serious adverse events (SAE) were registered at each study visit during the 3 vaccination cycles and boost cycles.
Time Frame: Change from baseline to end of Cycle 1 (3 months), end of Cycle 2 (8 months), end of Cycle 3 (13 months) and end of Boost Cycles (18 months to 23 months).
Population: After the end of a cycle, patients could have discontinue the study for personal reasons or PD. This is why the overall number of patients analyzed could change between cycles of each arm/group.
Measure: Mean (Standard Deviation); unit: Number of adverse events
Groups:
- 1.Melan-A ELA: 500 mcg Melan-A ELA analog peptide + 1 ml Montanide
- 2.Melan-A ELA + NY-ESO-1b(A) + MAGE-A10: 500 mcg Melan-A ELA analog peptide + 500 mcg NY-ESO-1b(A) analog peptide + 500 mcg MAGE-A10 peptide + 1 ml Montanide
- 3.Melan-A ELA + NY-ESO-1b(A) + MAGE-A10 + CpG: 500 mcg Melan-A ELA analog peptide + 500 mcg NY-ESO-1b(A) analog peptide + 500 mcg MAGE-A10 peptide + 1 ml Montanide + 2.5 mg CpG-7909/PF-3512676
- 4.Melan-A EAA/ELA + NY-ESO-1lp + MAGE-A10+ CpG: * If patient is HLA-A2 positive: 100 mcg Melan-A EAA native peptide (during first cycle) or 100 mcg ELA analog peptide (during other cycles) + 500 mcg NY-ESO-1lp long peptide + 100 mcg MAGE-A10 peptide + 1 ml Montanide (no Montanide during cycle 3) + 2.5 mg CpG-7909/PF-3512676
  * If patient is HLA-A2 negative: 500 mcg NY-ESO-1lp long peptide+ 1 ml Montanide (no Montanide during cycle 3) + 2.5 mg CpG-7909/PF-3512676
- 5.Melan-A EAA/ELA + NY-ESO-1lp + MAGE-A10+ CpG + IL-2: * If patient is HLA-A2 positive: 100 mcg Melan-A EAA native peptide (during first cycle) or 100 mcg ELA analog peptide (during other cycles) + 500 mcg NY-ESO-1lp long peptide + 100 mcg MAGE-A10 peptide + 1 ml Montanide (no Montanide during cycle 3) + 2.5 mg CpG-7909/PF-3512676 + low dose IL-2
  * If patient is HLA-A2 negative: 500 mcg NY-ESO-1lp long peptide+ 1 ml Montanide (no Montanide during cycle 3) + 2.5 mg CpG-7909/PF-3512676 + low dose IL-2
Arm/Group | 1.Melan-A ELA | 2.Melan-A ELA + NY-ESO-1b(A) + MAGE-A10 | 3.Melan-A ELA + NY-ESO-1b(A) + MAGE-A10 + CpG | 4.Melan-A EAA/ELA + NY-ESO-1lp + MAGE-A10+ CpG | 5.Melan-A EAA/ELA + NY-ESO-1lp + MAGE-A10+ CpG + IL-2
Number analyzed (Participants) | 10 | 5 | 5 | 10 | 9
Number of adverse events
  End of Cycle 1 | 13.40 (13.02) | 18.40 (5.86) | 23.80 (12.15) | 19.60 (8.15) | 31.75 (18.92)
  End of Cycle 2: number analyzed (Participants) | 9 | 4 | 4 | 9 | 5
  End of Cycle 2 | 10.44 (7.46) | 10.00 (7.62) | 20.25 (13.33) | 21.00 (12.30) | 16.80 (10.45)
  End of Cycle 3: number analyzed (Participants) | 5 | 3 | 4 | 6 | 2
  End of Cycle 3 | 6.20 (4.20) | 16.00 (9.74) | 21.25 (12.10) | 19.67 (12.92) | 20.50 (9.61)
  Boot cycles: number analyzed (Participants) | 3 | 3 | 3 | 1 | 0
  Boot cycles | 8.50 (6.54) | 9.00 (5.81) | 48.67 (53.87) | 50 (0.00) |

2. Primary Outcome: Fold Change From Baseline in ex Vivo Melan-A-specific CD8+ T Cells Frequency During the Vaccination Period
Description: Ex vivo frequency of Melan-A-specific CD8+ T cells was measured by multimer technique (tetramer assay) in a multicolor flow cytometry analysis.
  The fold change for each time point compared to baseline was calculated as: Melan-A-specific CD8+ T cell frequency at the time point/ Melan-A-specific CD8+ T cell frequency at baseline.
  Significant T cell response is defined by at least 2-fold change of Melan-A-specific CD8+ T cell frequency as compared to pre-immunotherapy.
Time Frame: Fold change from baseline in Melan-A-specific CD8+T-cells at the end of Cycle 1 (3 months), at the end of Cycle 2 (8 months), at the end of Cycle 3 (13 months) and if applicable at the end of Boost cycles (18 to 24 months).
Population: This test was only performed in patients HLA-A2 positive and Melan-A peptide positive (groups 1, 2 and 3, some patients from groups 4 and 5)
Measure: Mean (Standard Deviation); unit: Fold change of % Melan-A ELA+ CD8+ T
Groups:
- 2. Melan-A ELA + NY-ESO-1b(A) + MAGE-A10: 500 mcg Melan-A ELA analog peptide + 500 mcg NY-ESO-1b (A) analog peptide + 500 mcg Mage-A10 peptide + 1 ml Montanide
- 3. Melan-A ELA + NY-ESO-1b(A) + MAGE-A10 + CpG: 500 mcg Melan-A ELA analog peptide, 500 mcg + NY-ESO-1b(A) analog peptide + 500 mcg Mage-A10 peptide + 1 ml Montanide + 2.5 mg CpG-7909/PF-3512676
Arm/Group | 1. Melan-A ELA | 2. Melan-A ELA + NY-ESO-1b(A) + MAGE-A10 | 3. Melan-A ELA + NY-ESO-1b(A) + MAGE-A10 + CpG | 4. Melan-A EAA/ELA + NY-ESO-1lp + MAGE-A10+ CpG | 5. Melan-A EAA/ELA + NY-ESO-1lp + MAGE-A10+ CpG + IL-2
Number analyzed (Participants) | 10 | 5 | 5 | 5 | 2
Fold change of % Melan-A ELA+ CD8+ T
  Baseline | 0.03 (0.03) | 0.01 (0.01) | 0.08 (0.15) | 0.18 (0.29) | 0.04 (0.01)
  End of Cycle 1 | 0.08 (0.11) | 0.08 (0.08) | 0.37 (0.33) | 0.12 (0.16) | 0.05 (0.01)
  End of Cycle 2: number analyzed (Participants) | 8 | 3 | 4 | 3 | 1
  End of Cycle 2 | 0.07 (0.06) | 0.14 (0.12) | 0.34 (0.31) | 0.20 (0.22) | 0.26 (NA) — Only values for one patient
  End of Cycle 3: number analyzed (Participants) | 5 | 3 | 4 | 2 | 0
  End of Cycle 3 | 0.10 (0.07) | 0.08 (0.07) | 0.85 (1.36) | 0.09 (0.09) |
  End of Boost Cycles: number analyzed (Participants) | 3 | 3 | 3 | 0 | 0
  End of Boost Cycles | 0.04 (0.03) | 0.09 (0.06) | 2.66 (2.72) |  |

3. Primary Outcome: Fold Change From Baseline in ex Vivo Frequency of Melan-A-specific IFN-γ-secreting CD8+ T Cells During the Vaccination Period
Description: Ex vivo frequency of Melan-A-specific CD8+ T cells producing IFN-γ (Interferon-gamma) was measured through the Enzyme-Linked Immunosorbent Spot (ELISpot) assay.
  The fold change for each time point compared to baseline was calculated as: Melan-A-specific IFN-γ-secreting CD8+ T cell frequency at the time point/ Melan-A-specific IFN-γ-secreting CD8+ T cell frequency at baseline.
Time Frame: Fold change from baseline in Melan-A-specific IFN-γ-secreting CD8+T-cells frequency at the end of Cycle 1 (3 months), at the end of Cycle 2 (8 months), at the end of Cycle 3 (13 months) and if applicable at the end of Boost cycles (18 to 24 months)
Population: This test was only done in patients HLA-A2 positive and Melan-A peptide positive (groups 1, 2 and 3, some patients from groups 4 and 5)
Measure: Mean (Standard Deviation); unit: Fold change of % IFN-γ+ MelanA+ CD8+ T
Groups:
- Melan-A EAA/ELA + NY-ESO-1lp + MAGE-A10+ CpG + IL-2: * If patient is HLA-A2 positive: 100 mcg Melan-A EAA native peptide (during first cycle) or 100 mcg ELA analog peptide (during other cycles) + 500 mcg NY-ESO-1lp long peptide + 100 mcg MAGE-A10 peptide + 1 ml Montanide (no Montanide during cycle 3) + 2.5 mg CpG-7909/PF-3512676 + low dose IL-2
  * If patient is HLA-A2 negative: 500 mcg NY-ESO-1lp long peptide+ 1 ml Montanide (no Montanide during cycle 3) + 2.5 mg CpG-7909/PF-3512676 + low dose IL-2
Arm/Group | 1. Melan-A ELA | 2. Melan-A ELA + NY-ESO-1b(A) + MAGE-A10 | 3. Melan-A ELA + NY-ESO-1b(A) + MAGE-A10 + CpG | 4. Melan-A EAA/ELA + NY-ESO-1lp + MAGE-A10+ CpG | Melan-A EAA/ELA + NY-ESO-1lp + MAGE-A10+ CpG + IL-2
Number analyzed (Participants) | 10 | 5 | 5 | 5 | 1
Fold change of % IFN-γ+ MelanA+ CD8+ T
  Baseline | 0.001 (0.002) | 0.004 (0.006) | 0.065 (0.129) | 0.008 (0.012) | 0.150 (NA) — Only one patient analyzed
  End of Cycle 1 | 0 (0.003) | 0.015 (0.025) | 0.157 (0.458) | 0.018 (0.023) | 1.00 (NA) — Only one patient analyzed
  End of Cycle 2: number analyzed (Participants) | 8 | 3 | 4 | 3 | 0
  End of Cycle 2 | -0.003 (0.009) | 0.006 (0.006) | 0.015 (0.014) | 0.013 (0.011) |
  End of Cycle 3: number analyzed (Participants) | 6 | 3 | 4 | 1 | 0
  End of Cycle 3 | 0.010 (0.025) | 0.008 (0.003) | 0.068 (0.061) | -0.051 (NA) — Only one patient analyzed |
  End of Boost Cycles: number analyzed (Participants) | 3 | 3 | 3 | 0 | 0
  End of Boost Cycles | 0.027 (0.060) | 0.005 (0.005) | 0.380 (0.309) |  |

4. Primary Outcome: Fold Change From Baseline in ex Vivo Frequency of NY-ESO-1-specific CD8+ T Cells During the Vaccination Period
Description: Ex vivo frequency of NY-ESO-1-specific CD8+ T cells was measured by multimer technique (tetramer assay) in a multicolor flow cytometry analysis.
  The fold change for each time point compared to baseline was calculated as: NY-ESO-1-specific CD8+ T cell frequency at the time point/ NY-ESO-1-specific CD8+ T cell frequency at baseline.
Time Frame: Fold change from baseline in NY-ESO-1-specific CD8+T-cells at the end of Cycle 1 (3 months), at the end of Cycle 2 (8 months), at the end of Cycle 3 (13 months) and if applicable at the end of Boost cycles (18 to 24 months)
Population: This test was only done in patients HLA-A2 positive and NY-ESO-1 peptide positive (groups 2 and 3)
Measure: Mean (Standard Deviation); unit: Fold change of % NY-ESO-1+ CD8+ T cells
Arm/Group | 1. Melan-A ELA | 2. Melan-A ELA + NY-ESO-1b(A) + MAGE-A10 | 3. Melan-A ELA + NY-ESO-1b(A) + MAGE-A10 + CpG | 4. Melan-A EAA/ELA + NY-ESO-1lp + MAGE-A10+ CpG | 5. Melan-A EAA/ELA + NY-ESO-1lp + MAGE-A10+ CpG + IL-2
Number analyzed (Participants) | 0 | 5 | 5 | 0 | 0
Fold change of % NY-ESO-1+ CD8+ T cells
  Baseline |  | 0.69 (1.54) | 0.01 (0.02) |  |
  End of Cycle 1 |  | 0.96 (2.64) | 0.21 (0.28) |  |
  End of Cycle 2: number analyzed (Participants) | 0 | 3 | 4 | 0 | 0
  End of Cycle 2 |  | 2.37 (4.37) | 0.19 (0.23) |  |
  End of Cycle 3: number analyzed (Participants) | 0 | 3 | 4 | 0 | 0
  End of Cycle 3 |  | 2.64 (3.55) | 0.16 (0.24) |  |
  End of Boost Cycles: number analyzed (Participants) | 0 | 3 | 3 | 0 | 0
  End of Boost Cycles |  | 1.40 (2.40) | 0.1 (0.08) |  |

5. Primary Outcome: Fold Change From Baseline in ex Vivo Frequency of NY-ESO-1-specific IFN-γ-secreting CD8+ T Cells During the Vaccination Period
Description: Ex vivo frequency of NY-ESO-1-specific CD8+ T cells producing IFN-γ (Interferon-gamma) was measured through the Enzyme-Linked Immunosorbent Spot (ELISpot) assay.
  The fold change for each time point compared to baseline was calculated as: NY-ESO-1-specific IFN-γ-secreting CD8+ T cell frequency at the time point/ NY-ESO-1-specific IFN-γ-secreting CD8+ T cell frequency at baseline.
Time Frame: Fold change from baseline in NY-ESO-1-specific IFN-γ-secreting CD8+T-cells frequency at the end of Cycle 1 (3 months), at the end of Cycle 2 (8 months), at the end of Cycle 3 (13 months) and if applicable at the end of Boost cycles (18 to 24 months)
Population: This test was only done in patients HLA-A2 positive (groups 1, 2 and 3, some patients from groups 4 and 5)
Measure: Mean (Standard Deviation); unit: % of spots from NYESO1 specific CD8 cell
Arm/Group | 1. Melan-A ELA | 2. Melan-A ELA + NY-ESO-1b(A) + MAGE-A10 | 3. Melan-A ELA + NY-ESO-1b(A) + MAGE-A10 + CpG | 4. Melan-A EAA/ELA + NY-ESO-1lp + MAGE-A10+ CpG | 5. Melan-A EAA/ELA + NY-ESO-1lp + MAGE-A10+ CpG + IL-2
Number analyzed (Participants) | 10 | 5 | 5 | 5 | 1
% of spots from NYESO1 specific CD8 cell
  Baseline | 0.004 (0.01) | 0.218 (0.484) | 0.001 (0.001) | 0.010 (0.005) | 0.050 (NA) — Only values from one patient
  End of Cycle 1 | -0.001 (0.002) | 0.237 (0.491) | 0.004 (0.006) | 0.001 (0.005) | 0.030 (NA) — Only values from one patient
  End of Cycle 2: number analyzed (Participants) | 8 | 3 | 4 | 3 | 0
  End of Cycle 2 | 0.002 (0.004) | 0.378 (0.589) | -0.004 (0.040) | -0.003 (0.009) |
  End of Cycle 3: number analyzed (Participants) | 6 | 3 | 4 | 1 | 0
  End of Cycle 3 | -0.001 (0.008) | 0.538 (0.665) | -0.002 (0.065) | -0.111 (NA) — Only values from one patient |
  End of Boost Cycles: number analyzed (Participants) | 3 | 3 | 3 | 0 | 0
  End of Boost Cycles | -0.008 (0.011) | 0.045 (0.088) | 0.096 (0.121) |  |

6. Primary Outcome: Fold Change From Baseline in ex Vivo Frequency of MAGE-A10-specific CD8+ T Cells During the Vaccination Period
Description: Ex vivo frequency of MAGE-A10-specific CD8+ T cells was measured by multimer technique (tetramer assay) in a multicolor flow cytometry analysis.
  The fold change for each time point compared to baseline was calculated as: MAGE-A10-specific CD8+ T cell frequency at the time point/ MAGE-A10-specific CD8+ T cell frequency at baseline.
Time Frame: Fold change from baseline in MAGE-A10-specific CD8+T-cells at the end of Cycle 1 (3 months), at the end of Cycle 2 (8 months), at the end of Cycle 3 (13 months) and if applicable at the end of Boost cycles (18 to 24 months)
Population: This test was only done in patients MAGE-A10 positive and HLA-A2 positive (groups 2 and 3, some patients from groups 4 and 5)
Measure: Mean (Standard Deviation); unit: Fold change of % MAGE-A10+ CD8+ T cells
Arm/Group | 1. Melan-A ELA | 2. Melan-A ELA + NY-ESO-1b(A) + MAGE-A10 | 3. Melan-A ELA + NY-ESO-1b(A) + MAGE-A10 + CpG | 4. Melan-A EAA/ELA + NY-ESO-1lp + MAGE-A10+ CpG | 5. Melan-A EAA/ELA + NY-ESO-1lp + MAGE-A10+ CpG + IL-2
Number analyzed (Participants) | 0 | 5 | 5 | 5 | 2
Fold change of % MAGE-A10+ CD8+ T cells
  Baseline |  | 0 (0) | 0 (0) | 0 (0) | 0.04 (0.01)
  End of Cycle 1 |  | 0.03 (0.03) | 0.03 (0.02) | 0.01 (0.01) | 0.05 (0.01)
  End of Cycle 2: number analyzed (Participants) | 0 | 3 | 4 | 3 | 1
  End of Cycle 2 |  | 0.03 (0.02) | 0.05 (0.05) | 0.03 (0.03) | 0.26 (NA) — Only values from one patient
  End of Cycle 3: number analyzed (Participants) | 0 | 3 | 4 | 3 | 0
  End of Cycle 3 |  | 0.02 (0.01) | 0.03 (0.02) | 0.01 (0.01) |
  End of Boost Cycles: number analyzed (Participants) | 0 | 3 | 3 | 0 | 0
  End of Boost Cycles |  | 0.02 (0.02) | 0.07 (0.07) |  |

7. Primary Outcome: Fold Change From Baseline in ex Vivo Frequency of MAGE-A10-specific IFN-γ-secreting CD8+ T Cells During the Vaccination Period
Description: Ex vivo frequency of MAGE-A10-specific CD8+ T cells producing IFN-γ (Interferon-gamma) was measured through the Enzyme-Linked Immunosorbent Spot (ELISpot) assay.
  The fold change for each time point compared to baseline was calculated as: MAGE-A10-specific IFN-γ-secreting CD8+ T cell frequency at the time point/ MAGE-A10-specific IFN-γ-secreting CD8+ T cell frequency at baseline.
Time Frame: Fold change from baseline in MAGE-A10-specific IFN-γ-secreting CD8+T-cells frequency at the end of Cycle 1 (3 months), at the end of Cycle 2 (8 months), at the end of Cycle 3 (13 months) and if applicable at the end of Boost cycles (18 to 24 months)
Population: This test was only done in patients HLA-A2 positive (groups 1, 2 and 3, some patients from groups 4 and 5)
Measure: Mean (Standard Deviation); unit: Fold change of % IFN-γ+ MAGE-A10+ CD8+ T
Arm/Group | 1. Melan-A ELA | 2. Melan-A ELA + NY-ESO-1b(A) + MAGE-A10 | 3. Melan-A ELA + NY-ESO-1b(A) + MAGE-A10 + CpG | 4. Melan-A EAA/ELA + NY-ESO-1lp + MAGE-A10+ CpG | 5. Melan-A EAA/ELA + NY-ESO-1lp + MAGE-A10+ CpG + IL-2
Number analyzed (Participants) | 10 | 5 | 5 | 5 | 1
Fold change of % IFN-γ+ MAGE-A10+ CD8+ T
  Baseline | 0.001 (0.002) | 0.003 (0.006) | 0.014 (0.026) | 0 (0.005) | 0.09 (NA) — Only the value of one patient
  End of Cycle 1 | 0 (0.003) | 0.034 (0.079) | 0.004 (0.005) | 0.004 (0.005) | 0.120 (NA) — Only the value of one patient
  End of Cycle 2: number analyzed (Participants) | 8 | 3 | 4 | 3 | 0
  End of Cycle 2 | 0 (0.002) | 0.043 (0.076) | -0.006 (0.012) | 0.003 (0.002) |
  End of Cycle 3: number analyzed (Participants) | 6 | 3 | 4 | 1 | 0
  End of Cycle 3 | 0.015 (0.025) | 0.127 (0.154) | -0.016 (0.051) | -0.089 (NA) — Only the value of one patient |
  End of Boost Cycles: number analyzed (Participants) | 3 | 3 | 3 | 0 | 0
  End of Boost Cycles | -0.001 (0.020) | 0.004 (0.002) | 0.027 (0.044) |  |

8. Primary Outcome: Percentage of in Vitro Stimulated NY-ESO-1 Lp-specific IFN-γ/TNF-α -Secreting CD4+ T Cells During the Vaccination Period
Description: For each patient, total CD4+ T-cells were stimulated in the presence of peptide NY-ESO-1 long peptide (lp). After 10 days, cell cultures were challenged for 4h with the peptide or left unchallenged. The activation of NY-ESO-1 long peptide (lp)-specific CD4+ T cells were analyzed in vitro by Intracellular Cytokine Staining (ICS) via detection of IFN-γ (Interferon-gamma) and TNF-α (Tumor Necrosis Factor-alpha) producing cells.
Time Frame: Percentage of NY-ESO-1 lp-specific IFN-γ/TNF-α -secreting CD4+ T-cells at the end of Cycle 1 (3 months), at the end of Cycle 2 (8 months), at the end of Cycle 3 (13 months) and if applicable at the end of Boost cycles (18 to 24 months)
Population: Patients vaccinated with the NY-ESO-1 lp (groups 4 and 5). One patient of the group 5 received only one vaccine and thus was not included in the analysis of the immune response (the minimum dose required for immune response evaluation was 2 vaccines).
Measure: Mean (Standard Deviation); unit: % of NY-ESO-1 lp specific CD4+ T cells
Arm/Group | 1. Melan-A ELA | 2. Melan-A ELA + NY-ESO-1b(A) + MAGE-A10 | 3. Melan-A ELA + NY-ESO-1b(A) + MAGE-A10 + CpG | 4. Melan-A EAA/ELA + NY-ESO-1lp + MAGE-A10+ CpG | 5. Melan-A EAA/ELA + NY-ESO-1lp + MAGE-A10+ CpG + IL-2
Number analyzed (Participants) | 0 | 0 | 0 | 10 | 8
% of NY-ESO-1 lp specific CD4+ T cells
  NY-ESO-1lp T cells producing IFN-γ at baseline |  |  |  | 0.12 (0.21) | 071 (1.30)
  NY-ESO-1lp T cells producing TNF-α at baseline |  |  |  | 0.20 (0.36) | 1.05 (1.65)
  NY-ESO-1lp T cells producing IFN-γ _end of cycle 1 |  |  |  | 2.86 (4.94) | 16.24 (9.73)
  NY-ESO-1lp T cells producing TNF-α_ end of cycle 1 |  |  |  | 5.31 (3.83) | 23.69 (12.22)
  NY-ESO-1lp T cells IFN-γ_end of cycle 2: number analyzed (Participants) | 0 | 0 | 0 | 9 | 5
  NY-ESO-1lp T cells IFN-γ_end of cycle 2 |  |  |  | 1.81 (3.26) | 7.31 (4.74)
  NY-ESO-1lp T cells producing TNF-α _end of cycle 2: number analyzed (Participants) | 0 | 0 | 0 | 9 | 5
  NY-ESO-1lp T cells producing TNF-α _end of cycle 2 |  |  |  | 6.02 (5.79) | 17.10 (7.90)
  NY-ESO-1lp T cells IFN-γ _end of cycle 3: number analyzed (Participants) | 0 | 0 | 0 | 6 | 1
  NY-ESO-1lp T cells IFN-γ _end of cycle 3 |  |  |  | 7.02 (14.01) | 0.52 (NA) — Only one value from this group
  NY-ESO-1lp T cells producing TNF-α _end of cycle 3: number analyzed (Participants) | 0 | 0 | 0 | 6 | 1
  NY-ESO-1lp T cells producing TNF-α _end of cycle 3 |  |  |  | 10.00 (15.75) | 1.69 (NA) — Only one value from this group
  NY-ESO-1lp T producing IFN-γ _end of boost cycles: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0
  NY-ESO-1lp T producing IFN-γ _end of boost cycles |  |  |  | 19.47 (NA) — Only one value from this group |
  NY-ESO-1lp T producing TNF-α_end of boost cycles: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0
  NY-ESO-1lp T producing TNF-α_end of boost cycles |  |  |  | 21.11 (NA) — Only one value from this group |

9. Primary Outcome: Percentage of in Vitro Stimulated NY-ESO-1 Lp-specific IFN-γ/TNFα -Secreting CD8+ T Cells During the Vaccination Period
Description: For each patient, total CD8+ T cells were stimulated in the presence of peptide NY-ESO-1 long peptide (lp). After 10 days, cell cultures were challenged for 4h with the peptide or left unchallenged. The activation of NY-ESO-1 long peptide (lp)-specific CD8+ T cells were analyzed in vitro by Intracellular Cytokine Staining (ICS) via detection of IFN-γ (Interferon-gamma) and TNF-α (Tumor Necrosis Factor-alpha) producing cells.
Time Frame: Percentage of NY-ESO-1 lp-specific IFN-γ/TNF-α -secreting CD8+ T cells at the end of Cycle 1 (3 months), at the end of Cycle 2 (8 months), at the end of Cycle 3 (13 months) and if applicable at the end of Boost cycles (18 to 24 months)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: % of NY-ESO-1 lp specific CD8+ T cells
Arm/Group | 1. Melan-A ELA | 2. Melan-A ELA + NY-ESO-1b(A) + MAGE-A10 | 3. Melan-A ELA + NY-ESO-1b(A) + MAGE-A10 + CpG | 4. Melan-A EAA/ELA + NY-ESO-1lp + MAGE-A10+ CpG | 5. Melan-A EAA/ELA + NY-ESO-1lp + MAGE-A10+ CpG + IL-2
Number analyzed (Participants) | 0 | 0 | 0 | 10 | 8
% of NY-ESO-1 lp specific CD8+ T cells
  NY-ESO-1lp T cells producing IFN-γ at baseline |  |  |  | 0.03 (0.08) | 0.12 (0.17)
  NY-ESO-1lp T cells producing TNF-α at baseline |  |  |  | 0.02 (0.04) | 0.15 (0.26)
  NY-ESO-1lp T cells producing IFN-γ_end of cycle 1 |  |  |  | 0.88 (1.96) | 7.21 (8.40)
  NY-ESO-1lp T cells producing TNF-α_end of cycle 1 |  |  |  | 1.04 (2.08) | 7.74 (8.17)
  NY-ESO-1lp T cells producing IFN-γ_end of cycle 2: number analyzed (Participants) | 0 | 0 | 0 | 9 | 5
  NY-ESO-1lp T cells producing IFN-γ_end of cycle 2 |  |  |  | 0.34 (0.46) | 5.38 (6.69)
  NY-ESO-1lp T cells producing TNF-α_end of cycle 2: number analyzed (Participants) | 0 | 0 | 0 | 9 | 5
  NY-ESO-1lp T cells producing TNF-α_end of cycle 2 |  |  |  | 2.18 (3.48) | 4.21 (4.60)
  NY-ESO-1lp T cells producing IFN-γ_end of cycle 3: number analyzed (Participants) | 0 | 0 | 0 | 6 | 1
  NY-ESO-1lp T cells producing IFN-γ_end of cycle 3 |  |  |  | 0.93 (1.81) | 6.58 (NA) — Only one value for this group
  NY-ESO-1lp T cells producing TNF-α_end of cycle 3: number analyzed (Participants) | 0 | 0 | 0 | 6 | 1
  NY-ESO-1lp T cells producing TNF-α_end of cycle 3 |  |  |  | 1.01 (1.74) | 9.02 (NA) — Only one value for this group
  NY-ESO-1lp T producing IFN-γ_end of boost cycles: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0
  NY-ESO-1lp T producing IFN-γ_end of boost cycles |  |  |  | 0.22 (NA) — Only one value for this group |
  NY-ESO-1lp T producing TNF-α_end of boost cycles: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0
  NY-ESO-1lp T producing TNF-α_end of boost cycles |  |  |  | 0.36 (NA) — Only one value for this group |

10. Secondary Outcome: Disease Status Assessment During the Vaccination Period
Description: The disease status was assessed by computed tomography (CT) or positron emission tomography (PET)/CT at baseline and after the fourth vaccination of each cycle. During the "booster vaccines" period, imagery examinations were performed every 3 months for patients with measurable disease and every 6 months for patients with non measurable disease.
  The tumor response was assessed according to the classification World Health Organization (WHO) 1979 and defined as:
  * No Evidence of Disease (NED)
  * Stable disease (SD): Change in size of all measurable lesions (the sum of the products of the greatest and perpendicular parameters), of less than a 25% increase or 25% decrease from baseline for at least 4 weeks, without appearance of new lesions or progression of any lesion.
  * Progressing disease (PD): Appearance of new tumors, or increase in size of any measurable tumor by at least 25% of the sum of the product of the greatest and perpendicular diameter.
Time Frame: Disease status at baseline, after cycle 1 (3 months), after cycle 2 (8 months), after cycle 3 (13 months) and if applicable after boost cycles (16 months, 19 months or 22 months)
Population: Some patients discontinued treatment for either personal reasons or progressing disease. This is why from one cycle to other could be a decrease in the number of patients in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | 1. Melan-A ELA | 2. Melan-A ELA + NY-ESO-1b(A) + MAGE-A10 | 3. Melan-A ELA + NY-ESO-1b(A) + MAGE-A10 + CpG | 4. Melan-A EAA/ELA + NY-ESO-1lp + MAGE-A10+ CpG | 5. Melan-A EAA/ELA + NY-ESO-1lp + MAGE-A10+ CpG + IL-2
Number analyzed (Participants) | 10 | 5 | 5 | 10 | 9
Participants
  Baseline: Patients with No Evidence of Disease | 7 | 2 | 4 | 7 | 9
  Baseline: Patients with Stable Disease | 1 | 0 | 0 | 0 | 0
  Baseline: Patients with Progressing Disease | 2 | 3 | 1 | 3 | 0
  End of Cycle 1: Patients with No Evidence of Disease | 7 | 3 | 4 | 6 | 7
  End of Cycle 1: Patients with Stable Disease | 1 | 0 | 0 | 0 | 0
  End of Cycle 1: Patients with Progressing Disease | 2 | 2 | 1 | 4 | 2
  End of Cycle 2: number analyzed (Participants) | 9 | 4 | 4 | 9 | 5
  End of Cycle 2: Patients with No Evidence of Disease | 7 | 3 | 3 | 5 | 2
  End of Cycle 2: Patients with Stable Disease | 0 | 0 | 0 | 0 | 0
  End of Cycle 2: Patients with Progressing Disease | 2 | 1 | 1 | 4 | 3
  End of Cycle 3: number analyzed (Participants) | 6 | 3 | 4 | 6 | 2
  End of Cycle 3: Patients with No Evidence of Disease | 5 | 3 | 2 | 4 | 2
  End of Cycle 3: Patients with Stable Disease | 0 | 0 | 0 | 0 | 0
  End of Cycle 3: Patients with Progressing Disease | 1 | 0 | 2 | 2 | 0
  End of Boost Cycles: number analyzed (Participants) | 2 | 3 | 3 | 1 | 0
  End of Boost Cycles: Patients with No Evidence of Disease | 1 | 1 | 0 | 1 | 0
  End of Boost Cycles: Patients with Stable Disease | 0 | 0 | 0 | 0 | 0
  End of Boost Cycles: Patients with Progressing Disease | 1 | 2 | 3 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events (AE) were collected during the whole study period, from the first vaccination visit (V1, Day 0) to the last vaccination visit (V12) of the cycle 3 of vaccination (13 months) and if applicable during the boost periods (18 months to 23 months) therefore the adverse events were collected for 13 months if patients completed 3 cycles of vaccination and for 18 months to 23 months depending if patients received boost vaccinations.
Description: Adverse events (AE) that were expected (prelisted AE) and non expected (non prelisted AE), according to the Investigator's Brochure of the different vaccine components, were recorded during each visit from the first vaccination until the-end of the third cycle. During the "booster vaccinations" period, any AE were recorded the day of the vaccination and 7 days later. All AE were collected irrespective of their frequency, their severity and relationship to the study drug.
Arm/Group | 1. Melan-A ELA | 2. Melan-A ELA + NY-ESO-1b(A) + MAGE-A10 | 3. Melan-A ELA + NY-ESO-1b(A) + MAGE-A10 + CpG | 4. Melan-A EAA/ELA + NY-ESO-1lp + MAGE-A10+ CpG | 5. Melan-A EAA/ELA + NY-ESO-1lp + MAGE-A10+ CpG + IL-2
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/5 | 0/5 | 0/10 | 0/9
Serious Adverse Events (participants affected / at risk) | 1/10 | 1/5 | 1/5 | 3/10 | 2/9
Other Adverse Events (participants affected / at risk) | 10/10 | 5/5 | 5/5 | 10/10 | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1. Melan-A ELA (N=10) | 2. Melan-A ELA + NY-ESO-1b(A) + MAGE-A10 (N=5) | 3. Melan-A ELA + NY-ESO-1b(A) + MAGE-A10 + CpG (N=5) | 4. Melan-A EAA/ELA + NY-ESO-1lp + MAGE-A10+ CpG (N=10) | 5. Melan-A EAA/ELA + NY-ESO-1lp + MAGE-A10+ CpG + IL-2 (N=9)
Nephrectomy (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal colic (Renal and urinary disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Pulmonary granuloma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Post procedural infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Regional chemotherapy (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dehydration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Confusional state/ Dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1. Melan-A ELA (N=10) | 2. Melan-A ELA + NY-ESO-1b(A) + MAGE-A10 (N=5) | 3. Melan-A ELA + NY-ESO-1b(A) + MAGE-A10 + CpG (N=5) | 4. Melan-A EAA/ELA + NY-ESO-1lp + MAGE-A10+ CpG (N=10) | 5. Melan-A EAA/ELA + NY-ESO-1lp + MAGE-A10+ CpG + IL-2 (N=9)
Injection site erythema (Skin and subcutaneous tissue disorders) | 7 (24) | 5 (38) | 5 (72) | 9 (70) | 9 (63) — Local Reactions
Injection site induration (Skin and subcutaneous tissue disorders) | 9 (55) | 5 (44) | 5 (70) | 10 (73) | 9 (51) — Local Reactions
Injection site Pain (Skin and subcutaneous tissue disorders) | 6 (16) | 4 (21) | 5 (47) | 10 (73) | 7 (42) — Local Reactions
Injection site recall reaction (Skin and subcutaneous tissue disorders) | 4 (7) | 2 (5) | 2 (2) | 5 (10) | 4 (9) — Local Reactions
Injection site Warmth (Skin and subcutaneous tissue disorders) | 4 (8) | 1 (13) | 4 (44) | 8 (56) | 6 (30) — Local Reactions
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (3) | 2 (9) | 4 (13) | 5 (19) — Prelisted Systemic Reactions
Asthenia (General disorders) | 3 (4) | 0 (0) | 0 (0) | 2 (6) | 4 (13) — Prelisted Systemic Reactions
Chills (General disorders) | 2 (3) | 2 (2) | 3 (16) | 7 (32) | 5 (13) — Prelisted Systemic Reactions
Fever (General disorders) | 2 (10) | 0 (0) | 3 (16) | 7 (26) | 3 (5) — Prelisted Systemic Reactions
Headache (Nervous system disorders) | 2 (4) | 3 (8) | 3 (15) | 7 (44) | 5 (19) — Prelisted Systemic Reactions
influenza-like illness (General disorders) | 1 (1) | 1 (1) | 4 (32) | 3 (4) | 2 (2) — Prelisted Systemic Reactions
Malaise (General disorders) | 1 (1) | 2 (2) | 4 (14) | 4 (11) | 1 (2) — Prelisted Systemic Reactions
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (6) | 1 (1) | 2 (10) | 6 (39) | 5 (25) — Prelisted Systemic Reactions
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (3) | 3 (12) | 6 (14) | 4 (12) — Prelisted Systemic Reactions
Pruritus (General disorders) | 4 (7) | 0 (0) | 1 (1) | 2 (2) | 4 (9) — Prelisted Systemic Reactions
Ear Discharge (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Non-Prelisted Reactions
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Non-Prelisted Reactions
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Non-Prelisted Reactions
Chronic otitis (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Non-Prelisted Reactions
Gynecomastia (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Non-Prelisted Reactions
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Non-Prelisted Reactions
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) — Non-Prelisted Reactions
Chest pain-cardiac (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Non-Prelisted Reactions
Myocardial ischemia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Non-Prelisted Reactions
Heart murmurs (Cardiac disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Non-Prelisted Reactions
Tachycardi (Cardiac disorders) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (1) — Non-Prelisted Reactions
Ventricular arythmia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Non-Prelisted Reactions
Cardiac shock (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Non-Prelisted Reactions
Decrease visual field (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Non-Prelisted Reactions
Eye irritation (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) — Non-Prelisted Reactions
Visual troubles (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Non-Prelisted Reactions
Eyelid oedema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Non-Prelisted Reactions
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Non-Prelisted Reactions
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) — Non-Prelisted Reactions
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Non-Prelisted Reactions
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 2 (2) — Non-Prelisted Reactions
Diarrhoea (Gastrointestinal disorders) | 2 (3) | 1 (2) | 0 (0) | 0 (0) | 5 (11) — Non-Prelisted Reactions
Colitic lesions (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Non-Prelisted Reactions
Gastrointestinal disorders (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Non-Prelisted Reactions
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Non-Prelisted Reactions
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Non-Prelisted Reactions
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Non-Prelisted Reactions
Glossitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) — Non-Prelisted Reactions
Odynosphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Non-Prelisted Reactions
Oral Aphtha (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Non-Prelisted Reactions
Gastroenteritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Non-Prelisted Reactions
Left hypoesthesia mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Non-Prelisted Reactions
Sensitivity of teeth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) — Non-Prelisted Reactions
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Non-Prelisted Reactions
Discomfort (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) — Non-Prelisted Reactions
fatigue (Gastrointestinal disorders) | 5 (6) | 3 (4) | 1 (4) | 4 (4) | 5 (6) — Non-Prelisted Reactions
pain (General disorders) | 3 (3) | 1 (2) | 1 (1) | 1 (1) | 0 (0) — Non-Prelisted Reactions
Oedema (General disorders) | 3 (4) | 1 (1) | 0 (0) | 0 (0) | 1 (1) — Non-Prelisted Reactions
Localized oedema (General disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) — Non-Prelisted Reactions
Infusion site extravasation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) — Non-Prelisted Reactions
Throat glar (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Non-Prelisted Reactions
Immune system disorders (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Non-Prelisted Reactions
Granuloma (Immune system disorders) | 0 (0) | 3 (8) | 0 (0) | 0 (0) | 0 (0) — Non-Prelisted Reactions
Hepatic cysts (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Non-Prelisted Reactions
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Non-Prelisted Reactions
Cystitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Non-Prelisted Reactions
Erysipelas (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Non-Prelisted Reactions
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) — Non-Prelisted Reactions
Herpes labialis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Non-Prelisted Reactions
Infection inguinal scar (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Non-Prelisted Reactions
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) — Non-Prelisted Reactions
Post-operative infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Non-Prelisted Reactions
Prostate infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Non-Prelisted Reactions
Rhinitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) — Non-Prelisted Reactions
Bronchial infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Non-Prelisted Reactions
Laryngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Non-Prelisted Reactions
Mucosal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Non-Prelisted Reactions
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Non-Prelisted Reactions
Pharyngitis (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Non-Prelisted Reactions
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Non-Prelisted Reactions
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) — Non-Prelisted Reactions
Lund injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Non-Prelisted Reactions
Anemia (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Non-Prelisted Reactions
Elevated CK (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) — Non-Prelisted Reactions
Karnofsky scale worsened (Investigations) | 5 (8) | 0 (0) | 0 (0) | 6 (9) | 0 (0) — Non-Prelisted Reactions
Elevated liver values (due to Dafalgan) (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Non-Prelisted Reactions
Platelet count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Non-Prelisted Reactions
Lymphopenia (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Non-Prelisted Reactions
GGT increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) — Non-Prelisted Reactions
High ALP level (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Non-Prelisted Reactions
High LDH level (Investigations) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) — Non-Prelisted Reactions
High C-Reactive Protein (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Non-Prelisted Reactions
Increased of liver enzymes values (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Non-Prelisted Reactions
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) — Non-Prelisted Reactions
Weight increased (Investigations) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) — Non-Prelisted Reactions
Weight loss (Investigations) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Non-Prelisted Reactions
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 2 (4) — Non-Prelisted Reactions
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Non-Prelisted Reactions
Dehydratation (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 | 0 (0) | 0 (0) — Non-Prelisted Reactions
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) — Non-Prelisted Reactions
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Non-Prelisted Reactions
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Non-Prelisted Reactions
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Non-Prelisted Reactions
Axillary pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Non-Prelisted Reactions
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0) | 2 (4) | 0 (0) — Non-Prelisted Reactions
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (10) | 1 (1) | 3 (11) | 0 (0) | 0 (0) — Non-Prelisted Reactions
Metastasis skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 3 (7) | 1 (2) | 0 (0) | 1 (1) — Non-Prelisted Reactions
Prostatic hyperplasia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Non-Prelisted Reactions
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Non-Prelisted Reactions
Inguinal adenophathy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 2 (2) | 0 (0) | 3 (4) | 0 (0) — Non-Prelisted Reactions
Axillary adenopathy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (3) | 1 (1) | 0 (0) — Non-Prelisted Reactions
Mediastinal adenopathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Non-Prelisted Reactions
Cysts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Non-Prelisted Reactions
Black nodule on scar (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Non-Prelisted Reactions
Increased renal kystis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Non-Prelisted Reactions
Liver hemangiomas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Non-Prelisted Reactions
Neoplasms benign, malignant and unspecified-subcutaneous nodule (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (9) | 2 (4) | 2 (5) | 0 (0) | 0 (0) — Non-Prelisted Reactions
Ataxia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Non-Prelisted Reactions
Brain oedema (Nervous system disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) — Non-Prelisted Reactions
Carpal tunnel symdrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Non-Prelisted Reactions
Convulsion (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Non-Prelisted Reactions
Paresthesi (Nervous system disorders) | 3 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Non-Prelisted Reactions
Dysarthrya (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Non-Prelisted Reactions
Dysesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Non-Prelisted Reactions
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Non-Prelisted Reactions
Dysphasia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Non-Prelisted Reactions
Migraine (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Non-Prelisted Reactions
Sleeping disorders (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Non-Prelisted Reactions
Spasticity (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Non-Prelisted Reactions
Tremor (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Non-Prelisted Reactions
Vasovagal reaction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) — Non-Prelisted Reactions
Nervous Descompensation (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Non-Prelisted Reactions
Sensitivity impairment (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) — Non-Prelisted Reactions
Ischemia cerebrovascular (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Non-Prelisted Reactions
Temporal lobe (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Non-Prelisted Reactions
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) — Non-Prelisted Reactions
Agitation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Non-Prelisted Reactions
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Non-Prelisted Reactions
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) — Non-Prelisted Reactions
Mood alteration (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Non-Prelisted Reactions
Anuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Non-Prelisted Reactions
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Non-Prelisted Reactions
Renal colic (Renal and urinary disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) — Non-Prelisted Reactions
Urinary frequency (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Non-Prelisted Reactions
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Non-Prelisted Reactions
Amenorrhoea (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Non-Prelisted Reactions
Irregular menstruation (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Non-Prelisted Reactions
Menorrhagia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Non-Prelisted Reactions
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Non-Prelisted Reactions
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) — Non-Prelisted Reactions
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Non-Prelisted Reactions
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) — Non-Prelisted Reactions
Chronic cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) — Non-Prelisted Reactions
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0) — Non-Prelisted Reactions
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) — Non-Prelisted Reactions
Induration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) — Non-Prelisted Reactions
Hyperhydrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Non-Prelisted Reactions
Itching/Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Non-Prelisted Reactions
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Non-Prelisted Reactions
Dermohypodermitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Non-Prelisted Reactions
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Non-Prelisted Reactions
Keratosis lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) — Non-Prelisted Reactions
Macular skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Non-Prelisted Reactions
Skin scab (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Non-Prelisted Reactions
Ingrown toe nail (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Non-Prelisted Reactions
Difficult cicatrization (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) — Non-Prelisted Reactions
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) — Non-Prelisted Reactions
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) — Non-Prelisted Reactions
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) — Non-Prelisted Reactions
Skin depigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Non-Prelisted Reactions
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Non-Prelisted Reactions
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Non-Prelisted Reactions
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Non-Prelisted Reactions
Scar (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Non-Prelisted Reactions
Pain scar (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Non-Prelisted Reactions
Haematoma post-biopsy (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Non-Prelisted Reactions
Motor skills decrease after brain surgery (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Non-Prelisted Reactions
Lymph node dissection (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Non-Prelisted Reactions
Metastasis resection (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Non-Prelisted Reactions
Post-operative pain (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) — Non-Prelisted Reactions
Post-operative arythmia (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Non-Prelisted Reactions
Punch-biopsy previous injection site (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Non-Prelisted Reactions
Broken foot toe (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Non-Prelisted Reactions
Hypertension (Vascular disorders) | 1 (2) | 0 (0) | 2 (2) | 1 (1) | 0 (0) — Non-Prelisted Reactions
Hypotension (Vascular disorders) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Non-Prelisted Reactions
Haematoma (Vascular disorders) | 3 (3) | 0 (0) | 2 (3) | 1 (2) | 3 (4) — Non-Prelisted Reactions
Hot Flush (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Non-Prelisted Reactions
Lymphedema (Vascular disorders) | 2 (2) | 2 (2) | 1 (2) | 0 (0) | 1 (1) — Non-Prelisted Reactions
Varix (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Non-Prelisted Reactions

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No